CLINICAL TRIAL: NCT01855893
Title: Effectiveness of the Auto-acupressure for Diminishing Neck Pain of Benign Origin
Brief Title: Auto-acupressure: Effectiveness for Diminishing Neck Pain of Benign Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Susana Calvo Trujillo, PhD, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12/00203
Record Dates: First submitted 2013-05-08; First posted 2013-05-17 (Estimated); Last update posted 2017-06-09 (Actual); Status verified 2017-03

CONDITIONS: Neck Pain
Keywords: Neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Auto-acupressure (Experimental): Patients will receive instructions about how to apply auto-acupressure once in a day during one week by their health care professionals.This technique will be complementary to the conventional treatment.
  Interventions: Other: Auto-acupressure
- Conventional treatment (Other): Conventional treatment consist of: 7 days with paracetamol 1g /8 hours and/ or ibuprofen 400mg/ 8 hours, and tetrazepam 50 mg/ 12 hours
  Interventions: Other: Conventional treatment

INTERVENTIONS:
Other: Auto-acupressure — Patients will receive instructions about how to apply auto-acupressure once in a day during one week by their health care professionals.This technique will be complementary to the conventional treatment.
  Arms: Auto-acupressure
Other: Conventional treatment — Conventional treatment consist of: 7 days with paracetamol 1g /8 hours and/ or ibuprofen 400mg/ 8 hours, and tetrazepam 50 mg/ 12 hours
  Arms: Conventional treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the auto-acupressure (digital pressure in points of acupuncture) added to the conventional treatment.

DETAILED DESCRIPTION:
OBJECTIVE: To evaluate the effectiveness of the digital pressure in points of acupuncture added to the conventional treatment for diminishing the pain in patients with cervicalgia of benign origin.

MATERIAL AND METHODS: Pragmatic controlled randomized clinical trial. Patients with diagnosis of cervicalgia of benign origin will include. They will be randomly assigned to receive just conventional treatment or this plus auto-acupressure.

The professionals will once receive instruction in the Centres of Health by an experienced acupuncture professional that will supervise, in a workshop, the right application of the technique, that will consist of the application of manoeuvres of auto-acupressure by the own patient during periods of 10 minutes, once in a day during one week. The pain intensity will be evaluated by means of a millimetric scale of 10 cm (0 represents the pain absence, 10 the maximum imaginable pain, Numerical Scale Rating). The pain will be measured in the inclusion and days 1, 3, 7, 30 and 90. The sample size has been calculated to detect a minimum difference of 1.5 points (DS 2) in the scale of the pain in day 7, which implies the recruitment of, at least, 80 patients by group (if losses don't exceed 20%). Also the perception of the quality of life (euroQol-5D) and the functional capacity with the scale of Oswestry will be evaluated, at the beginning, and days 3, 7, 30 and 90. The measures in each point between the group will be compared control and intervention. The evolution of the repeated measures will compare between groups with a generalized estimating equation (GEE) model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who come to consultation of Primary Care for neck pain without structural hurt or irradiation, with muscular contraction and functional and postural limitation.

Exclusion Criteria:

* Injuries of skin (dermatitis, burns, sores, skin cancer) in the zone to massaging
* Structural injuries (bony fractures or injuries of muscles and tendons) in the zone to massaging
* Hemorrhage or tendency to suffer hemorrhage
* Chronic, serious diseases
* Malignant diseases and marked physical deterioration
* Psychiatric disorders
* Sensitive alterations
* Treatment with drugs of second or third level of the scale of the WHO which difficult to estimate changes for auto-acupressure
* No sign the informed consent
* Difficulty of reading comprehension or visual alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Ninety days
  The pain intensity will be evaluated by means of a millimetric scale of 10 cm (Numerical Rating Scale)

SECONDARY OUTCOMES:
Perception of quality of life | Ninety days
  The perception of quality of life will be evaluated by EuroQol 5D

CONTACTS AND LOCATIONS:
Overall Officials: Susana Calvo-Trujillo, MD, Principal Investigator — Gerencia Atención Primaria. Madrid
Locations (1):
- Gerencia de Atención Primaria, Madrid, Spain

REFERENCES:
- [Derived] Susana CT, Maria TML, Pilar DS, Maria MMT, Pilar MS, Valentin MG; group EDIDO-CUH. Effectiveness of self-applied acupressure for cervical pain of benign origin (EDIDO-CUH): a randomized controlled clinical trial. Acupunct Med. 2021 Oct;39(5):441-451. doi: 10.1177/0964528420961398. Epub 2020 Dec 6. PMID 33280397